CLINICAL TRIAL: NCT05015400
Title: Female Urogenital Nutrition- Health Study
Acronym: FUN-Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Kaila Vento, Principal Investigator, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00014289
Record Dates: First submitted 2021-08-09; First posted 2021-08-20 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Bacterial Urinary Tract Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluid Increase (Experimental): The increased fluid intervention arm will begin on day 2 after the onset of bleeding (day 1) of their phase 1 menses through day 5. For the increased fluid intake intervention, participants will a) consume an additional 64 oz (1.89 L) of plain water only on top of habitual fluid intake and b) aim to at least urinate 5 times per day.
  Interventions: Other: Plain Water
- Fluid Habitual (No Intervention): The fluid habitual non-intervention arm will a) maintain normal fluid intake volume and beverage choices and a) urination frequency.

INTERVENTIONS:
Other: Plain Water — To increase water fluid intake, an additional 1.89 L, during phase 1 of the menstrual cycle (days 1-5).
  Arms: Fluid Increase

SUMMARY:
The purpose of this study is to assess nutrition and urinary tract bacterial activity during menstruation of approximately 15 female university Reserve Officer Training Corps (ROTC) cadets and Phoenix area police officers, firefighters, and military veterans.

DETAILED DESCRIPTION:
Urinary tract infections (UTIs) disrupt tactical service women's obligations and health, which increases sexual transmitted infections (STIs), HPV, and cervical cancer risk if left untreated. Females are more susceptible to UTIs due to their unique anatomical features and hormone fluctuations affecting vaginal flora. During phase 1 of the menstrual cycle (i.e., onset of bleeding, menstrual cycle days 1-5), estrogen levels significantly decrease and inhibit the growth of lactobacilli (good bacteria), which is essential in warding off bad bacteria and infections, particularly UTIs. The uropathogenic bacterial growth in phase 1 could be heightened in phase 2 of the menstrual cycle (i.e., leading to ovulation), as increases in estrogen favors bacteria adhesion and arginine vasopressin (AVP) release that stimulates fluid retention, leading to less volume flow in the urinary tract. To reduce UTI onset, it is recommended to frequently urinate with sufficient urine void volume to facilitate washing out harmful bacteria from the urethra and bladder. While menstruating, increased fluid consumption to support urination frequency and void volume may be critical, as the urinary tract is more predisposed to infections, and the effects of estrogen on bacterial adhesion and AVP release in phase 2 could continue uropathogenic growth.

Question(s) 1: Are premenopausal tactical service women's current hydration status and behaviors (i.e., fluid intake and urination) sufficient? How many premenopausal tactical service women have a UTI history?

Question 2: Will increasing daily water intake of identified underhydrated tactical service women reduce uropathogenic bacterial activity during the first part (i.e., onset of bleeding through day 5) of the menstrual cycle?

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-34 years of age or older (premenopausal)
* Have a 21-35-day menstrual cycle
* No changes in hormonal contraceptives within the last three months
* No current UTI symptoms
* Sexual activity and inactivity

Exclusion Criteria:

* Males
* Under 18 years of age or over 34 years of age
* Pregnant or nursing
* Menstrual irregularities effecting having a menstrual cycle to be between 21-35 days
* Progesterone-only contraceptive use (combined estrogen-progesterone and non-hormonal IUDs are okay)
* Currently taking antibiotics
* On hormone replacement therapy
* Currently experiencing symptomatic vulvovaginitis
* Diagnosed with recurrent UTI
* Not volunteering to participate

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2021-09-05 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Uropathogenic Bacterial Activity | Change from Baseline Uropathogenic Bacterial Activity at 1 month
  Number of bacterial colonies and uropathogens found

SECONDARY OUTCOMES:
Hydration Status | Change from Baseline Hydration Status at 1 month
  Urine concentration via urine specific gravity

CONTACTS AND LOCATIONS:
Overall Officials: Kaila A Vento, PhD(c), Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication.